CLINICAL TRIAL: NCT07090395
Title: Severe Label Expansion for EVO Products Trial
Acronym: SLEEP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ProSomnus Sleep Technologies (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SP-005
Record Dates: First submitted 2025-06-23; First posted 2025-07-29 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Obstructive Sleep Apnea
Keywords: oral appliance therapy; mandibular advancement device; ProSomnus
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- EVO Sleep and Snore Device (Experimental)
  Interventions: Device: EVO Sleep and Snore Device

INTERVENTIONS:
Device: EVO Sleep and Snore Device — ProSomnus EVO Sleep and Snore Device mandibular advancement device

SUMMARY:
Title: Severe Label Expansion for EVO Positioner (SLEEP) Study Description: Single-arm study to determine the safety and effectiveness of treating severe obstructive sleep apnea using the EVO Sleep and Snore Device (ProSomnus Sleep Technologies, Pleasanton, CA).

Objectives: To determine the safety and effectiveness of the EVO Sleep and Snore Device in individuals with severe obstructive sleep apnea.

Endpoints: The primary effectiveness endpoint is the Sher criteria defined as a reduction of Apnea-Hypopnea Index (AHI) of at least 50% from the baseline value and a post-treatment AHI of less than 20 events/hour at 6 months following initiation of Oral Appliance Therapy (OAT) titration. AHI will be collected using HSAT at baseline and 6 months. The primary safety objective is to evaluate safety by summarizing all reported device and/or procedure related adverse events from the time the EVO device is introduced through 6 months. Study Population: A maximum of 49 individuals over the age of 18 years with severe obstructive sleep apnea will be enrolled.

Description of Sites/Facilities Enrolling Participants: The study will be conducted at up to four sites, up to two of which could be located outside of the US. Description of Study Device: The study device is the EVO Sleep and Snore Device (ProSomnus Sleep Technologies, Pleasanton, CA). The device is a mandibular repositioning device used to treat obstructive sleep apnea. The device is currently cleared for the treatment of mild and moderate OSA.

Study Duration: The time from when the study opens to enrollment until completion of data analyses is estimated to be 15 months.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female, aged 18-80 years (inclusive)
4. Diagnosed with uncomplicated severe OSA (AHI > 30 h-1); where uncomplicated is defined by the absence of:

   1. Conditions that place the patient at increased risk of non-obstructive sleep-disordered breathing (e.g., central sleep apnea, hypoventilation, and sleep-related hypoxemia [e.g., resulting from severe chronic obstructive, interstitial lung disease, or pulmonary hypertension]). Examples of such conditions include significant cardiopulmonary disease (congestive heart failure, recurrent atrial fibrillation, coronary artery disease, resistant hypertension), potential respiratory muscle weakness due to neuromuscular conditions, history of stroke, and chronic opiate medication use.
   2. Concern for significant non-respiratory sleep disorder(s) that require evaluation (e.g., disorders of central hypersomnolence, parasomnias, sleep-related movement disorders) or interfere with accuracy of HSAT (e.g., severe insomnia).
   3. Environmental or personal factors that preclude the adequate acquisition and interpretation of data from HSAT.
5. Body mass index (BMI) < 35 kg/m2
6. Absence of severe oxyhemoglobin desaturation during sleep, indicated by mean nocturnal SpO2 > 87%
7. Adequate mandibular range of motion
8. Adequate dentition

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Inability to breathe through the nose comfortably
2. Presence of > 25% CSA
3. Presence of positional OSA per Amsterdam Positional OSA Classification I definition
4. History of surgery intended to alter anatomy for the correction of OSA

   1. E.g., uvulopalatopharyngoplasty (UPPP), maxillomandibular advancement (MMA), tongue/hyoid suspension, slow maxillary expansion
   2. History of surgery intended to restore normal anatomy, such as tonsillectomy, adenoidectomy, septoplasty, or polypectomy, is permitted.
5. Presence of hypoglossal nerve stimulation device (active or inactive)
6. Use of CPAP or OAT within the two weeks prior to the baseline sleep study
7. History of OAT that has been confirmed to provide effective therapy within the two years prior to the baseline sleep study
8. Anticipated change in medical therapy during the study protocol that could alter OSA severity (e.g., weight loss surgery, weight loss drug, UPPP, MMA, tongue/hyoid suspension, etc.)
9. Loose teeth or advanced periodontal disease
10. History of temporomandibular joint disorder
11. Resistant hypertension, defined as inadequately controlled blood pressure despite therapy with

    ≥ 3 oral hypertensive agents
12. Use of pacemaker or other life-supporting device
13. Participation in other studies that could interfere with the study protocol
14. Pregnancy or lactation
15. In the opinion of the investigator, unsuitable for inclusion in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Sher responder rate endpoint | 6 months
  Proportion of participants who meet the Sher criteria at outcome, defined as a reduction of apnea-hypopnea index less than 20 events/hour and 50% or greater reduction from the baseline value.
Incidence of adverse events | 6 months
  Evaluation of safety by summarizing all reported device- and/or procedure-related adverse events from the time the EVO device is introduced through 6 months.

SECONDARY OUTCOMES:
Sleep apnea-specific hypoxic burden | 6 months
  Proportion of participants achieving a sleep apnea-specific hypoxic burden less than 60 %min/h at 6 months
Epworth Sleepiness Scale change from baseline | 6 months
  Change in Epworth Sleepiness Scale from baseline to 6 months. The Epworth Sleepiness Scale ranges from 0 to 24, with 0 being the lowest and 24 being the highest score indicating propensity for sleep.
Sher criteria responder rate point estimate | 6 months
  Responder rate point estimate for the Sher criteria post-titration and at 6 months
Severity classification change | 6 months
  OSA severity classification change from baseline to post-titration and 6 months
Apnea-hypopnea index change from baseline | 6 months
  Change in AHI, ODI and SASHB change from baseline to 6 months
Oxygen desaturation index change from baseline | 6 months
  Change in oxygen desaturation index from baseline to 6 months
Sleep apnea-specific hypoxic burden change from baseline | 6 months
  Change in sleep apnea-specific hypoxic burden from baseline to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Erin Mosca, PhD, Study Director — ProSomnus Sleep Technologies
Locations (1):
- Star Sleep and Wellness, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No